CLINICAL TRIAL: NCT06332339
Title: A First-in-human Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of 16055 NFL Delta Gly4 Env Protein Trimer and Trimer 4571 Combined With 3M-052-AF + Alum Adjuvant and Ad4-Env145NFL Viral Particles as Heterologous Prime-boost Regimens in Adult Participants Without HIV
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of 16055 NFL Delta Gly4 Env Protein Trimer and Trimer 4571 Combined With 3M-052-AF + Alum Adjuvant and Ad4-Env145NFL Viral Particles as Heterologous Prime-boost Regimens in Adult Participants Without HIV.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 313
Record Dates: First submitted 2024-02-21; First posted 2024-03-27 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: HIV

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment 1 (Experimental): 16055 NFL delta Gly4 trimer, 200 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate intramuscular (IM) injections (0.27 mL each) at months 0, 2, 4, 8, and 12.
  Interventions: Biological: 16055 NFL delta Gly4 trimer
- Treatment 2 (Experimental): 16055 NFL delta Gly4 trimer, 200 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.27 mL each) at months 0 and 2.
  Ad4-Env145NFL, 5 x 108 viral particles (vp) to be administered intranasally (IN) (0.07 mL into 1 nostril) at month 4.
  Trimer 4571, 100 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.2 mL each) at months 8 and 12.
  Interventions: Biological: 16055 NFL delta Gly4 trimer; Biological: Trimer 4571; Biological: Ad4-Env145NFL, 5 x 108 viral particles (vp)
- Treatment 3 (Experimental): 16055 NFL delta Gly4 trimer, 200 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.27 mL each) at months 0 and 2.
  Trimer 4571, 100 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.2 mL each) at month 4.
  Ad4-Env145NFL, 5 x 108 vp to be administered IN (0.07 mL into 1 nostril) at months 8 and 12.
  Interventions: Biological: 16055 NFL delta Gly4 trimer; Biological: Trimer 4571; Biological: Ad4-Env145NFL, 5 x 108 viral particles (vp)

INTERVENTIONS:
Biological: 16055 NFL delta Gly4 trimer — 200 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.27 mL each)
Biological: Trimer 4571 — 100 mcg admixed with 3M-052-AF, 5 mcg and Alum, 500 mcg to be administered as 2 separate IM injections (0.2 mL each)
  Arms: Treatment 2; Treatment 3
Biological: Ad4-Env145NFL, 5 x 108 viral particles (vp) — to be administered intranasally (IN) (0.07 mL into 1 nostril)
  Arms: Treatment 2; Treatment 3

SUMMARY:
The goal of this clinical trial is to test 16055 NFL delta Gly4 Env protein trimer and Trimer 4571 combined with 3M-052-AF + Alum adjuvant and Ad4-Env145NFL viral particles as heterologous prime-boost regimens in adult participants without HIV.

The main question[s] it aims to answer are:

* Are these vaccine regimens safe and well tolerated?
* Are the prime-boost vaccine regimens that include Ad4-Env145NFL and Trimer 4571 as heterologous boosts going contribute to the development of B-cell and antibody responses?

Participants will attend scheduled study visits to receive their vaccine and will record symptoms on a daily eDiary.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): Volunteer demonstrates an understanding of this study and completes a questionnaire prior to signing the informed consent form with verbal demonstration of understanding of questionnaire items that were answered incorrectly.
* 18 to 55 years old, inclusive, on day of enrollment.
* Available for clinic follow-up and willing to undergo study procedures through the last clinic visit.
* Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 313 PSRT are required prior to enrollment into HVTN 313
* In good general health according to the clinical judgment of the site investigator.
* Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
* Assessed by clinical staff as having a low likelihood of acquiring HIV per guidelines, agrees to discuss their potential for HIV acquisition, agrees to risk-reduction counseling, and agrees to avoid behaviors associated with a higher likelihood of acquiring HIV through the final study visit. Low likelihood may include persons stably taking pre-exposure prophylaxis (PrEP) as prescribed.
* Hemoglobin (Hgb):

  * ≥ 11.0 g/dL for volunteers who were assigned female sex at birth (AFAB)
  * ≥ 13.0 g/dL for volunteers who were assigned male sex at birth (AMAB) and for transgender men who have been on hormone therapy for more than 6 consecutive months
  * ≥ 12.0 g/dL for transgender women who have been on hormone therapy for more than 6 consecutive months
  * For transgender volunteers who have been on hormone therapy for less than 6 consecutive months, determine hemoglobin eligibility based on the sex assigned at birth.
* White blood cell (WBC) count = 2,500 to 12,000/mm³ (WBC over 12,000/mm³ is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
* Platelets = 125,000 to 550,000/mm³.
* Alanine aminotransferase (ALT) within the institutional normal range.
* Serum creatinine ≤ 1.1 x upper limit of normal (ULN) based on the institutional normal range.
* Serum calcium level of > 8.5 mg/dL (if the participant consented to have leukapheresis as a study procedure).
* Blood pressure (BP) in the range of 90 to < 140 mmHg systolic and 50 to < 90 mmHg diastolic.
* Negative HIV test results by one of the following options: For US volunteers:

  * US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA)
  * Chemiluminescent microparticle immunoassay (CMIA)
  * Two negative results on HIV rapid tests (one of which must be FDA-approved CMIA)
* Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV Abs are detected.
* Negative for Hepatitis B surface antigen.
* For AFAB or intersex at birth volunteers who are capable of becoming pregnant (hereafter referred to as "persons of pregnancy potential"):

  * Must agree to use effective means of birth control from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint (see Appendix H).
  * Must have a negative beta human chorionic gonadotropin (β-HCG) pregnancy test (urine or serum) on day of enrollment.
* AMAB or intersex at birth volunteers must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.
* AMAB volunteers must agree to consistently practice abstinence or another method of effective birth control during sexual intercourse with persons of pregnancy potential and must not donate sperm at least 21 days prior to each Ad4-Env145NFL vaccination through 28 days following each Ad4-Env145NFL vaccination.
* Willing to follow precautions as provided by the study team for preventing the spread of adenovirus in the community.

Inclusion criteria for contacts of Ad4-Env145NFL vaccinees:

* Able and willing to complete the informed consent process, including an Assessment of Understanding (AoU): Volunteer demonstrates an understanding of this study and completes a questionnaire prior to enrollment with verbal demonstration of understanding of questionnaire items that were answered incorrectly.
* Meets criteria of a household contact or intimate contact.

  * A household contact is someone who resides (ie, lives in the same house or apartment) with the potential vaccinee within the first 28 days following each Ad4-Env145NFL vaccination.
  * An intimate contact is defined as someone who engages in mouth-to-mouth kissing, sexual intercourse, or oral sex with the study participant within the first 28 days following each Ad4-Env145NFL vaccination.
* Available for clinic follow-up and willing to participate in study procedures through the last scheduled clinic visit for the observational cohort.
* Age ≥ 18 years old on the day of enrollment.

Exclusion Criteria:

* Volunteer who is breastfeeding or pregnant.
* Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT on a case-by-case basis.
* Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
* Previous or current recipient of an investigational HIV vaccine (previous placebo recipients are not excluded).
* Receipt of non-HIV experimental vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) emergency use listing (EUL).
* Congenital or acquired immunodeficiency, including systemic medication (includes oral, intramuscular, or intravenously administrated medications) use likely to impair immune response to vaccine in the opinion of the site investigator, such as systemic glucocorticoid use equal to or greater than prednisone 10 mg/day within 3 months prior to enrollment.
* Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
* Receipt of any live, attenuated, replicating vaccine within 4 weeks prior to enrollment or planned administration within 4 weeks after enrollment. Note for ACAM2000 vaccine for mpox (formerly known as Monkeypox): the vaccination scab must no longer be present and at least 4 weeks is required prior to enrollment.
* Receipt or planned receipt of any killed/subunit/inactivated/non-replicating vaccine within 2 weeks prior to enrollment or planned administration within 2 weeks after enrollment. This applies to Jynneos vaccine for mpox which is non- replicating.
* Initiation of antigen-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
* Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life greater than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
* History of serious reaction (e.g., hypersensitivity, anaphylaxis) to any related vaccine or component of the study-vaccine regimen.
* Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
* Idiopathic urticaria within the past year.
* Bleeding disorder diagnosed by a clinician which would make study procedures a contraindication.
* Seizure disorder; febrile seizures as a child or seizures secondary to alcohol withdrawal more than 5 years ago are not exclusionary.
* Asplenia or functional asplenia.
* Active duty and reserve US military personnel.
* Any other chronic or clinically significant condition that, in the clinical judgement of the investigator, would jeopardize the safety or rights of the study participant, including, but not limited to: clinically significant forms of substance use disorder or alcohol use disorder, serious psychiatric disorders, persons with any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has a potential for recurrence (excluding basal cell carcinoma).
* Asthma is excluded if the participant has ANY of the following:

  * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year, OR
  * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or co-existing conditions unrelated to asthma); OR
  * Uses a short-acting rescue inhaler more than 2 days/week for acute asthma symptoms (i.e., not for preventive treatment prior to athletic activity); OR
  * Uses medium-to-high-dose inhaled corticosteroids (greater than 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (i.e., with a long-acting beta agonist, OR
  * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
* A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Specific examples are listed in Appendix I (AESI index). Not exclusionary: mild psoriasis that does not require ongoing systemic treatment.
* Investigator concern for difficulty with venous access based upon clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.
* Individuals who expect to live in the same household with or provide care for any of the following, within 28 days following each of the third through fifth study vaccination timepoints:

  * An individual under 5 years of age
  * An individual who is immunocompromised, immunosuppressed, or has any condition which would place them at undue risk for complications of an adenoviral infection, per the investigator's judgement
  * A person who is currently pregnant or breastfeeding or planning a pregnancy during the period of study vaccination
* Individuals who are unable or unwilling to avoid intimate contact for at least 28 days following each Ad4-Env145NFL vaccination with individuals with any of the following:

  * Immunocompromised or immunosuppressed condition
  * Are currently pregnant or breastfeeding or planning a pregnancy during the period of study vaccination
  * Any condition which would place them at undue risk for complications of an adenoviral infection, per the investigator's judgement
* History of thrombosis with thrombocytopenia (TTS) or HIT with or without thrombosis.
* History of a medical condition, including use of intranasal steroids that compromises the integrity of the nasal/cerebrospinal fluid (CSF) barrier and poses undue risk for complications of the Ad4-Env145NFL IN vaccination, per investigator judgement.
* History of a surgical condition that compromises the integrity of the nasal/cerebrospinal fluid (CSF) barrier and poses undue risk for complications of the Ad4-Env145NFL IN vaccination, per investigator judgement.

Exclusion criteria for contacts of Ad4-Env145NFL vaccinees:

* Any condition that, in the investigator's judgment, places the participant at undue risk by participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-11-11 (Estimated); Study Completion 2026-11-11 (Estimated)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms | 2 weeks following any injection
  for a minimum of 14 days following receipt of intramuscular injections and intranasal administrations of study products.
Systemic reactogenicity signs and symptoms | 2 weeks following any injection
  for a minimum of 14 days following receipt of intramuscular injections and intranasal administrations of study products.
Number of adverse events (AEs) reported for 30 days after receipt of any study product | 30 days following any injection
Number of Serious Adverse Reactions (SAEs) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of Medically Attended Adverse Event (MAAEs) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of Adverse Events of Special Interest (AESIs) that are Potential Immune Mediated Medical Conditions (PIMMCs) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Number of Adverse Events (AEs) leading to early participant withdrawal or permanent discontinuation | 12 months following receipt of any study product
Occurrence of serum IgG binding antibodies to vaccine-matched HIV-1 Env trimers and specific epitopes (e.g., CD4 binding site, V2, base of trimer, etc) | Week 34 (following the 4th vaccine), Week 54 for Group 1, 2, and Week for Group 3 (following the 5th vaccine)
  Measured by binding antibody multiplex assay (BAMA) after the fourth and fifth vaccinations.
Magnitude of serum IgG binding antibodies to vaccine-matched HIV-1 Env trimers and specific epitopes (e.g., CD4 binding site, V2, base of trimer, etc.) | Week 34 (following the 4th vaccine), Week 54 for Group 1, 2, and Week for Group 3 (following the 5th vaccine)
  measured by binding antibody multiplex assay (BAMA) after the fourth and fifth vaccinations
Response Rate of serum IgG binding antibodies to vaccine-matched HIV-1 Env trimers and specific epitopes (e.g., CD4 binding site, V2, base of trimer, etc.) | Week 34 (following the 4th vaccine), Week 54 for Group 1, 2, and Week for Group 3 (following the 5th vaccine)
  measured by binding antibody multiplex assay (BAMA) after the fourth and fifth vaccinations

SECONDARY OUTCOMES:
Occurrence of serum antibody neutralization of the autologous pseudovirus HIV-1 strains (including vaccine-matched deglycosylated 16055, WT 16055, BG505, 1086) | 2 weeks after the second vaccination and following subsequent vaccinations
  as measured by the TZM-bl assay
Magnitude of serum antibody neutralization of the autologous pseudovirus HIV-1 strains (including vaccine-matched deglycosylated 16055, WT 16055, BG505, 1086) | 2 weeks after the second vaccination and following subsequent vaccinations
  as measured by the TZM-bl assay
Response Rate of serum antibody neutralization of the autologous pseudovirus HIV-1 strains (including vaccine-matched deglycosylated 16055, WT 16055, BG505, 1086) | 2 weeks after the second vaccination and following subsequent vaccinations
  as measured by the TZM-bl assay
Occurrence of serum antibody neutralization of HIV-1 strains | Through study completion, an average of 1 year
  as measured by TZM-bl assay to a panel of tier 1 and tier 2 HIV-1 strains
Magnitude of serum antibody neutralization of HIV-1 strains | Week 34 (following the 4th vaccine), Week 54 for Group 1, 2, and Week for Group 3 (following the 5th vaccine)
  as measured by TZM-bl assay to a panel of tier 1 and tier 2 HIV-1 strains
Response Rate of serum antibody neutralization of HIV-1 strains | Week 34 (following the 4th vaccine), Week 54 for Group 1, 2, and Week for Group 3 (following the 5th vaccine)
  as measured by TZM-bl assay to a panel of tier 1 and tier 2 HIV-1 strains
Flow cytometry analysis of the frequency of Env-specific IgG+ B cells | Week 34 (following the 4th vaccine), Week 54 (following the 5th vaccine)
Occurrence of serum IgG binding antibodies as measured by BAMA | 2 weeks after second and third vaccinations
Magnitude of serum IgG binding antibodies as measured by BAMA | 2 weeks after second and third vaccinations
Response Rate of serum IgG binding antibodies as measured by BAMA | 2 weeks after second and third vaccinations
Number of Isolation of CD4bs bnAb specific VH and VL alleles and characteristic mutations | Through study completion, an average of 1 year
  as measured by B-cell receptor (BCR) sequencing
Flow cytometry analysis of the frequency of Env-specific IgG+ B cells at 26 weeks and 52 weeks after the fifth vaccination | At 26 weeks and 52 weeks after the fifth vaccination
Occurrence of serum IgG binding antibodies | 26 weeks after the fifth vaccination
  as measured by BAMA
Magnitude of serum IgG binding antibodies | 26 weeks after the fifth vaccination
  as measured by BAMA
Response Rate of serum IgG binding antibodies | 26 weeks after the fifth vaccination
  as measured by BAMA
Occurrence of serum antibody neutralization to tier 2 HIV-1 strains | 26 weeks after the fifth vaccination
  as measured by the TZM-bl assay 26 weeks after the fifth vaccination
Magnitude of serum antibody neutralization to tier 2 HIV-1 strains | 26 weeks after the fifth vaccination
  as measured by the TZM-bl assay 26 weeks after the fifth vaccination
Response Rate of serum antibody neutralization to tier 2 HIV-1 strains | 26 weeks after the fifth vaccination
  As measured by the TZM-bl assay 26 weeks after the fifth vaccination.
Epitope specific response rates as measured by electron microscopy polyclonal epitope mapping (EMPEM) | Week 18 (following the 3rd vaccine), Week 34 (following the 4th vaccine) and Week 54 (following the 5th vaccine)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Alabama CRS, Birmingham, Alabama
  - The Hope Clinic of the Emory Vaccine Center CRS Site# 31440, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - University of Rochester HIV/AIDS CTU, Rochester, New York
  - University of Pennsylvania HIV Therapeutics and Prevention Clinical Trials Unit, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No